CLINICAL TRIAL: NCT06231836
Title: High-flow Nasal Oxygenation Versus Standard Oxygenation for Gastrointestinal Endoscopy With Sedation in Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMASU Master 763/2023
Record Dates: First submitted 2024-01-08; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Prevention of Intraoperative Hypoxia
MeSH Terms: interventions — Cannula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High flow nasal cannula group (Active Comparator)
  Interventions: Device: High flow nasal cannula (HFNO)
- Nasal cannula group (Active Comparator)
  Interventions: Device: nasal cannula

INTERVENTIONS:
Device: High flow nasal cannula (HFNO) — O2 is administered by HFNO with flow 70L/min and the FiO2 is set at 40%,
  Arms: High flow nasal cannula group
Device: nasal cannula — O2 is administered by nasal cannula at 6L/min
  Arms: Nasal cannula group

SUMMARY:
Hypoxaemia is a major complication during gastrointestinal endoscopy (GIE) procedures (upper/lower) when performed under deep sedation in the procedure room especially with a body mass index above 30 kg/m².

The objective of the present work is to compare the use of High-flow nasal oxygenation (HFNO) with Standard oxygen therapy (SOT) in obese patient undergoing GIE.

DETAILED DESCRIPTION:
• Pre-operative settings:

1. All patients will be subjected to full history taking and thorough physical examination.
2. Age, sex and American Society Association (ASA) physical status were recorded.
3. Preoperative investigations will be done to all patients including laboratory investigations.
4. Oxygen saturation (SpO2) is recorded in ambient air
5. preoperative monitoring including ECG, non-invasive blood pressure and SpO2 via pulse oximeter are displayed and recorded in each patient using standard anaesthesia monitors.
6. Arterial Blood Gase(ABG) are sampled on room air .

Intraoperative settings:

* According to ASA standard monitoring criteria (pulse oximeter, non-invasive blood pressure cuff and electrocardiogram) will be attached to all patients.
* All patients will be monitored for peripheral oxygen saturation, blood pressure, Electrocardiogram through the whole operation.
* Intravenous access will be applied under aseptic condition, SpO2 is recorded in ambient air.
* Preoxygenation with the oxygen device (face mask 10L/min) for 3 min before starting the induction.
* The induction is done by An initial bolus of propofol (0.5-1 mg/kg) is administered intravenously, followed by a repeated bolus (10-20 mg) according to the patient's condition, or a continuous propofol infusion (2-6 mg/kg/h, with an additional bolus administered as needed) The infusion rate is chosen according to the desired sedation depth and the patient risk profile .
* In group A(intervention group) : preoxygenation for 3 min ,then start induction .Once the eyelash reflex has disappeared O2 is administered by HFNO with flow 70L/min and the FiO2 is set at 40%,The decision to set the FiO2 at 40% was made to obtain a similar FiO2 in both groups and to reduce the risk of hyperoxia and hypercapnia.
* In group B(control group):preoxygenation for 3 min, after induction ,once the eyelash reflex has disappeared, O2 is administered by nasal cannula at 6L/min.
* The investigator- chose to set a similar initial FiO2 in both groups during preoxygenation and procedure not to disadvantage the SOT group, as similar FiO2 will allow to determine if the HFNO- induced Positive End Expiratory Pressure PEEP and dead space washout effects could be beneficial.
* During the procedure, in both groups, if deemed necessary, the investigator can raise the FiO2 or the gas flow in case of desaturation or for any reason.
* In case of major intolerance, HFNO or SOT can be stopped and replaced by any other oxygen therapy technique.
* Tracheal intubation is allowed if necessary. In every case, investigators have to record all events in the case report form.

Post-operative settings:

* At the end of the GIE, patients are transferred to the recovery room and the interventional period is over. HFNO is not used in the recovery room. In the recovery room, SOT is immediately applied to all patients until deemed unnecessary, according to our current practice.
* All patients are monitoring for one hour in the recovery room then transfer them to the ward and this is the end point of study.
* ABGs are sampled in the recovery to detect the risk of hypercapnia in our study.

ELIGIBILITY:
Inclusion Criteria:

* Obese patient with body mass index (BMI) >30
* Patients scheduled for GIE (upper and/or lower endoscopy), for which sedation with maintenance of spontaneous breathing is planned.
* Patients older than 18 years old.

Exclusion Criteria:

* Gastrointestinal endoscopy (GIE) performed in emergency.
* Necessity to intubate the patient for the procedure.
* Patient under oxygen therapy at home.
* Tracheostomised patient.
* Pregnancy.
* Patient not affiliated or excluded from social protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
occurence of hypoxia | during the procedure
  SpO2 <90%

SECONDARY OUTCOMES:
occurence of hypoxia | from recovery room admission till discharge up to one hour
  SpO2 ≤92%
The rate of modifications of oxygen flow in both groups and of the FiO2 in the HFNO group. | during the procedure
number of participants needed to use mask ventilation or to perform any airway intervention | during the procedure
number of participants needed non- invasive ventilation, laryngeal mask airway or for intubation | during the procedure
number of participants needed to stop the procedure | during the procedure
occurence of hypercapnia (end tidal carbon dioxide >40 millimeter mercury) | during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No